CLINICAL TRIAL: NCT06029400
Title: CT-based Myocardial Characterization
Brief Title: CT-based Myocardial Characterization (CTMyoC)
Acronym: CTMyoC
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Antonio Esposito, Professor, IRCCS San Raffaele
Other Study IDs: CTMyoC
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: The retrospective arm of the study will include 200 patients meeting the inclusion criteria who have received a cardiac CT from January 2013 to date of approval amendment. (2013 was chosen as starting year to retrieve CT and clinical date in order to have at least 5 years of follow-up per patients).
- Prospective cohort: The prospective arm of the study will include 2000 consecutive patients meeting the inclusion criteria, candidate to cardiac CT along the 7 years after date of approval.

SUMMARY:
The identification of myocardial fibrosis in term of myocardial scar and extracellular matrix remodelling assessed respectively with the technique of Late Gadolinium Enhancement (LGE) and with the quantification of the Extracellular Volume Fraction (ECV) in Cardiac Magnetic Resonance has been demonstrated to be crucial in the diagnosis of different cardiomyopathy and to be prognosticators of major cardiovascular adverse events [1-14].

For these reason CMR represent the gold standard for the non-invasive characterization of myocardial tissue in the clinical practice.

However, regardless of its indisputable clinical role, CMR has many limitations: 1) it does not allow to evaluate coronary arteries; 2) it is contraindicated in patients with cardiac devices, and in case of conditional device they may also significantly impair LGE assessability due to artefacts [19]); 2) has limited availability and it is time consuming, therefore it is difficult to perform in the acute setting also because of poor patient compliance; 3) it is not feasible in patients suffering from claustrophobia. Cardiac Computed Tomography (cCT) is the image of choice to non-invasively study coronary arteries, not assessable with CMR. Moreover the recent technological advancement has continuously increased the clinical indication to the evaluation of cardiac valve and fibrosis, with reduced acquisition time respect to CMR (few minutes vs 1 hour), radiation exposure and costs.

cCT has emerging as a possible alternative to CMR in the characterization of myocardial scar and extracellular volume fraction, with the advantage of a single shot evaluation of coronary arteries and myocardial tissue remodelling (scar, diffuse fibrosis, contractility..).In particular, several studies including some from our group, have demonstrated the clinical utility of myocardial tissue characterization with cCT in different clinical settings, such as myocardial infarction [20, 21], myocarditis [22], hypertrophic cardiomyopathy (HCM) [23], heart failure [24], ventricular tachycardia [25], and sarcoidosis [26]. Despite the interesting results, all these previous studies are limited on highly selected and small sample size. Moreover, any large study with long term follow-up is available in the setting of tissue characterization (myocardial scar and ECV) in cCT also as well as combined with a multiparametric approach (cardiac chamber morphofuntionality,contractility-strain, valve calcification, geometry, coronary atherosclerosis, myocardial perfusion, myocardial strain and texture) and no data are available about its prognostic impact. Aim of the study is to evaluate the potential of cCT in tissue characterization (myocardial scar and ECV) alone and associate to other CT imaging biomarker on a large population of patient clinically candidate to cardiac CT.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* no contraindication to cCT
* signed informed consent
* clinical indication to cCT for the following reason: stable angina, heart failure, atrial/ ventricular arrhythmias, acute chest pain with need of "triple-rule-out" scan, planning of valvular repair/substitution, structural and infiltrative cardiomyopathy, new onset ECG alteration, troponin increase.

Exclusion Criteria:

* age < 18 years
* pregnancy and/or breastfeeding
* contraindications to iodinated contrast agent administration or impaired renal function (eGFR ≤ 30 mL/min);
* inability to sustain a brief breath hold (5 seconds)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a monocentric observational study with a retrospective and a prospective arms.
  Patients will be recruited from the Radiology Department of our Institution (IRCCS Ospedale San Raffaele, Milan, Italy). Written informed consent will be obtained.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2032-10-12 (Estimated); Study Completion 2032-10-12 (Estimated)

PRIMARY OUTCOMES:
Composite outcome | 60 months
  first hospitalization for heart failure (HHF) or death (all-cause mortality).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mewton N, Liu CY, Croisille P, Bluemke D, Lima JA. Assessment of myocardial fibrosis with cardiovascular magnetic resonance. J Am Coll Cardiol. 2011 Feb 22;57(8):891-903. doi: 10.1016/j.jacc.2010.11.013. PMID 21329834
- [Background] Kuruvilla S, Adenaw N, Katwal AB, Lipinski MJ, Kramer CM, Salerno M. Late gadolinium enhancement on cardiac magnetic resonance predicts adverse cardiovascular outcomes in nonischemic cardiomyopathy: a systematic review and meta-analysis. Circ Cardiovasc Imaging. 2014 Mar;7(2):250-258. doi: 10.1161/CIRCIMAGING.113.001144. Epub 2013 Dec 20. PMID 24363358
- [Background] Mavrogeni S, Petrou E, Kolovou G, Theodorakis G, Iliodromitis E. Prediction of ventricular arrhythmias using cardiovascular magnetic resonance. Eur Heart J Cardiovasc Imaging. 2013 Jun;14(6):518-25. doi: 10.1093/ehjci/jes302. Epub 2013 Jan 16. PMID 23324829
- [Background] Weng Z, Yao J, Chan RH, He J, Yang X, Zhou Y, He Y. Prognostic Value of LGE-CMR in HCM: A Meta-Analysis. JACC Cardiovasc Imaging. 2016 Dec;9(12):1392-1402. doi: 10.1016/j.jcmg.2016.02.031. Epub 2016 Jul 20. PMID 27450876
- [Background] Haaf P, Garg P, Messroghli DR, Broadbent DA, Greenwood JP, Plein S. Cardiac T1 Mapping and Extracellular Volume (ECV) in clinical practice: a comprehensive review. J Cardiovasc Magn Reson. 2016 Nov 30;18(1):89. doi: 10.1186/s12968-016-0308-4. PMID 27899132
- [Background] Bulluck H, Hammond-Haley M, Fontana M, Knight DS, Sirker A, Herrey AS, Manisty C, Kellman P, Moon JC, Hausenloy DJ. Quantification of both the area-at-risk and acute myocardial infarct size in ST-segment elevation myocardial infarction using T1-mapping. J Cardiovasc Magn Reson. 2017 Aug 1;19(1):57. doi: 10.1186/s12968-017-0370-6. PMID 28764773
- [Background] Youn JC, Hong YJ, Lee HJ, Han K, Shim CY, Hong GR, Suh YJ, Hur J, Kim YJ, Choi BW, Kang SM. Contrast-enhanced T1 mapping-based extracellular volume fraction independently predicts clinical outcome in patients with non-ischemic dilated cardiomyopathy: a prospective cohort study. Eur Radiol. 2017 Sep;27(9):3924-3933. doi: 10.1007/s00330-017-4817-9. Epub 2017 Apr 24. PMID 28439651
- [Background] Ferreira VM, Piechnik SK, Dall'Armellina E, Karamitsos TD, Francis JM, Ntusi N, Holloway C, Choudhury RP, Kardos A, Robson MD, Friedrich MG, Neubauer S. T(1) mapping for the diagnosis of acute myocarditis using CMR: comparison to T2-weighted and late gadolinium enhanced imaging. JACC Cardiovasc Imaging. 2013 Oct;6(10):1048-1058. doi: 10.1016/j.jcmg.2013.03.008. Epub 2013 Sep 4. PMID 24011774
- [Background] Hinojar R, Varma N, Child N, Goodman B, Jabbour A, Yu CY, Gebker R, Doltra A, Kelle S, Khan S, Rogers T, Arroyo Ucar E, Cummins C, Carr-White G, Nagel E, Puntmann VO. T1 Mapping in Discrimination of Hypertrophic Phenotypes: Hypertensive Heart Disease and Hypertrophic Cardiomyopathy: Findings From the International T1 Multicenter Cardiovascular Magnetic Resonance Study. Circ Cardiovasc Imaging. 2015 Dec;8(12):e003285. doi: 10.1161/CIRCIMAGING.115.003285. PMID 26659373
- [Background] Puntmann VO, Isted A, Hinojar R, Foote L, Carr-White G, Nagel E. T1 and T2 Mapping in Recognition of Early Cardiac Involvement in Systemic Sarcoidosis. Radiology. 2017 Oct;285(1):63-72. doi: 10.1148/radiol.2017162732. Epub 2017 Apr 27. PMID 28448233
- [Background] Martinez-Naharro A, Kotecha T, Norrington K, Boldrini M, Rezk T, Quarta C, Treibel TA, Whelan CJ, Knight DS, Kellman P, Ruberg FL, Gillmore JD, Moon JC, Hawkins PN, Fontana M. Native T1 and Extracellular Volume in Transthyretin Amyloidosis. JACC Cardiovasc Imaging. 2019 May;12(5):810-819. doi: 10.1016/j.jcmg.2018.02.006. Epub 2018 Mar 14. PMID 29550324
- [Background] Karur GR, Robison S, Iwanochko RM, Morel CF, Crean AM, Thavendiranathan P, Nguyen ET, Mathur S, Wasim S, Hanneman K. Use of Myocardial T1 Mapping at 3.0 T to Differentiate Anderson-Fabry Disease from Hypertrophic Cardiomyopathy. Radiology. 2018 Aug;288(2):398-406. doi: 10.1148/radiol.2018172613. Epub 2018 Apr 24. PMID 29688154
- [Background] Neilan TG, Coelho-Filho OR, Shah RV, Feng JH, Pena-Herrera D, Mandry D, Pierre-Mongeon F, Heydari B, Francis SA, Moslehi J, Kwong RY, Jerosch-Herold M. Myocardial extracellular volume by cardiac magnetic resonance imaging in patients treated with anthracycline-based chemotherapy. Am J Cardiol. 2013 Mar 1;111(5):717-22. doi: 10.1016/j.amjcard.2012.11.022. Epub 2012 Dec 8. PMID 23228924
- [Background] Treibel TA, Fridman Y, Bering P, Sayeed A, Maanja M, Frojdh F, Niklasson L, Olausson E, Wong TC, Kellman P, Miller CA, Moon JC, Ugander M, Schelbert EB. Extracellular Volume Associates With Outcomes More Strongly Than Native or Post-Contrast Myocardial T1. JACC Cardiovasc Imaging. 2020 Jan;13(1 Pt 1):44-54. doi: 10.1016/j.jcmg.2019.03.017. Epub 2019 May 15. PMID 31103587
- [Background] Barone-Rochette G, Pierard S, De Meester de Ravenstein C, Seldrum S, Melchior J, Maes F, Pouleur AC, Vancraeynest D, Pasquet A, Vanoverschelde JL, Gerber BL. Prognostic significance of LGE by CMR in aortic stenosis patients undergoing valve replacement. J Am Coll Cardiol. 2014 Jul 15;64(2):144-54. doi: 10.1016/j.jacc.2014.02.612. PMID 25011718
- [Background] Chin CWL, Everett RJ, Kwiecinski J, Vesey AT, Yeung E, Esson G, Jenkins W, Koo M, Mirsadraee S, White AC, Japp AG, Prasad SK, Semple S, Newby DE, Dweck MR. Myocardial Fibrosis and Cardiac Decompensation in Aortic Stenosis. JACC Cardiovasc Imaging. 2017 Nov;10(11):1320-1333. doi: 10.1016/j.jcmg.2016.10.007. Epub 2016 Dec 21. PMID 28017384
- [Background] Chaikriangkrai K, Lopez-Mattei JC, Lawrie G, Ibrahim H, Quinones MA, Zoghbi W, Little SH, Shah DJ. Prognostic value of delayed enhancement cardiac magnetic resonance imaging in mitral valve repair. Ann Thorac Surg. 2014 Nov;98(5):1557-63. doi: 10.1016/j.athoracsur.2014.06.049. Epub 2014 Sep 18. PMID 25240782
- [Background] Steen H, Madadi-Schroeder M, Lehrke S, Lossnitzer D, Giannitsis E, Katus HA. Staged cardiovascular magnetic resonance for differential diagnosis of troponin T positive patients with low likelihood for acute coronary syndrome. J Cardiovasc Magn Reson. 2010 Sep 14;12(1):51. doi: 10.1186/1532-429X-12-51. PMID 20840783
- [Background] Dickfeld T, Tian J, Ahmad G, Jimenez A, Turgeman A, Kuk R, Peters M, Saliaris A, Saba M, Shorofsky S, Jeudy J. MRI-Guided ventricular tachycardia ablation: integration of late gadolinium-enhanced 3D scar in patients with implantable cardioverter-defibrillators. Circ Arrhythm Electrophysiol. 2011 Apr;4(2):172-84. doi: 10.1161/CIRCEP.110.958744. Epub 2011 Jan 26. PMID 21270103
- [Background] Tanabe Y, Kido T, Kurata A, Kouchi T, Fukuyama N, Yokoi T, Uetani T, Yamashita N, Miyagawa M, Mochizuki T. Late iodine enhancement computed tomography with image subtraction for assessment of myocardial infarction. Eur Radiol. 2018 Mar;28(3):1285-1292. doi: 10.1007/s00330-017-5048-9. Epub 2017 Sep 19. PMID 28929333
- [Background] Rodriguez-Granillo GA. Delayed enhancement cardiac computed tomography for the assessment of myocardial infarction: from bench to bedside. Cardiovasc Diagn Ther. 2017 Apr;7(2):159-170. doi: 10.21037/cdt.2017.03.16. PMID 28540211
- [Background] Bouleti C, Baudry G, Iung B, Arangalage D, Abtan J, Ducrocq G, Steg PG, Vahanian A, Henry-Feugeas MC, Pasi N, Chillon S, Pitocco F, Laissy JP, Ou P. Usefulness of Late Iodine Enhancement on Spectral CT in Acute Myocarditis. JACC Cardiovasc Imaging. 2017 Jul;10(7):826-827. doi: 10.1016/j.jcmg.2016.09.013. Epub 2016 Dec 21. No abstract available. PMID 28017385
- [Background] Zhao L, Ma X, Delano MC, Jiang T, Zhang C, Liu Y, Zhang Z. Assessment of myocardial fibrosis and coronary arteries in hypertrophic cardiomyopathy using combined arterial and delayed enhanced CT: comparison with MR and coronary angiography. Eur Radiol. 2013 Apr;23(4):1034-43. doi: 10.1007/s00330-012-2674-0. Epub 2012 Oct 14. PMID 23064716
- [Background] Ohta Y, Kitao S, Yunaga H, Fujii S, Mukai N, Yamamoto K, Ogawa T. Myocardial Delayed Enhancement CT for the Evaluation of Heart Failure: Comparison to MRI. Radiology. 2018 Sep;288(3):682-691. doi: 10.1148/radiol.2018172523. Epub 2018 Jul 10. PMID 29989514
- [Background] Esposito A, Palmisano A, Antunes S, Maccabelli G, Colantoni C, Rancoita PMV, Baratto F, Di Serio C, Rizzo G, De Cobelli F, Della Bella P, Del Maschio A. Cardiac CT With Delayed Enhancement in the Characterization of Ventricular Tachycardia Structural Substrate: Relationship Between CT-Segmented Scar and Electro-Anatomic Mapping. JACC Cardiovasc Imaging. 2016 Jul;9(7):822-832. doi: 10.1016/j.jcmg.2015.10.024. Epub 2016 Feb 17. PMID 26897692
- [Background] Aikawa T, Oyama-Manabe N, Naya M, Ohira H, Sugimoto A, Tsujino I, Obara M, Manabe O, Kudo K, Tsutsui H, Tamaki N. Delayed contrast-enhanced computed tomography in patients with known or suspected cardiac sarcoidosis: A feasibility study. Eur Radiol. 2017 Oct;27(10):4054-4063. doi: 10.1007/s00330-017-4824-x. Epub 2017 Apr 5. PMID 28382537
- [Background] Nacif MS, Kawel N, Lee JJ, Chen X, Yao J, Zavodni A, Sibley CT, Lima JA, Liu S, Bluemke DA. Interstitial myocardial fibrosis assessed as extracellular volume fraction with low-radiation-dose cardiac CT. Radiology. 2012 Sep;264(3):876-83. doi: 10.1148/radiol.12112458. Epub 2012 Jul 6. PMID 22771879
- [Background] Marwan M, Achenbach S, Korosoglou G, Schmermund A, Schneider S, Bruder O, Hausleiter J, Schroeder S, Barth S, Kerber S, Leber A, Moshage W, Senges J. German cardiac CT registry: indications, procedural data and clinical consequences in 7061 patients undergoing cardiac computed tomography. Int J Cardiovasc Imaging. 2018 May;34(5):807-819. doi: 10.1007/s10554-017-1282-0. Epub 2017 Dec 1. PMID 29197025
- [Background] Knuuti J, Bengel F, Bax JJ, Kaufmann PA, Le Guludec D, Perrone Filardi P, Marcassa C, Ajmone Marsan N, Achenbach S, Kitsiou A, Flotats A, Eeckhout E, Minn H, Hesse B. Risks and benefits of cardiac imaging: an analysis of risks related to imaging for coronary artery disease. Eur Heart J. 2014 Mar;35(10):633-8. doi: 10.1093/eurheartj/eht512. Epub 2013 Dec 29. No abstract available. PMID 24375074
- [Background] Esposito A, Palmisano A, Barbera M, Vignale D, Benedetti G, Spoladore R, Ancona MB, Giannini F, Oppizzi M, Del Maschio A, De Cobelli F. Cardiac Computed Tomography in Troponin-Positive Chest Pain: Sometimes the Answer Lies in the Late Iodine Enhancement or Extracellular Volume Fraction Map. JACC Cardiovasc Imaging. 2019 Apr;12(4):745-748. doi: 10.1016/j.jcmg.2018.08.013. Epub 2018 Oct 17. No abstract available. PMID 30343092
- [Background] Vignale D, Palmisano A, Gnasso C, Margonato D, Romagnolo D, Barbieri S, Ingallina G, Stella S, Ancona MB, Montorfano M, Maisano F, Agricola E, Esposito A. Extracellular volume fraction (ECV) derived from pre-operative computed tomography predicts prognosis in patients undergoing transcatheter aortic valve implantation (TAVI). Eur Heart J Cardiovasc Imaging. 2023 Jun 21;24(7):887-896. doi: 10.1093/ehjci/jead040. PMID 36916015